CLINICAL TRIAL: NCT03336853
Title: A New Approach for Controlling Hemostasis During Canal Treatment: a Randomized Controlled Study
Brief Title: A New Approach for Controlling Hemostasis During Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Riccardo Pace (Other)
Responsible Party: Sponsor-Investigator, Dr Riccardo Pace, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Organization: Azienda Ospedaliero-Universitaria Careggi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: endo 2-2017
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Blood Contamination of Root Canal During Endodontic Therapy

STUDY DESIGN:
Intervention Model Description: single center, participants and data analyst blind, two-arm, randomized, placebo controlled clinical trial study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HybenX ® (Experimental): 1 cc of mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%) for 20 sec
  Interventions: Device: HybenX
- Control (Placebo Comparator): 5 cc of sterile saline water for 20 sec
  Interventions: Other: Placebo control

INTERVENTIONS:
Device: HybenX — The material was introduced inside the root canal using the pre-dosed syringe for 20 seconds with a sterile paper point with and up and down movement up to the working length.
  Finally, the canal was rinsed with sterile water using a syringe with a side-vented 30 G needle 1 mm shorter than the working length.
  A second sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect the presence of blood and the millimeters of blood inside the root canal was measured again according the previous criteria.
  Arms: HybenX ®
Other: Placebo control — The root canal was irrigated with sterile saline water with a syringe and a side-vented 30G needle activated for 20 seconds with a sterile paper point with and up and down movement up to the working length to ensure a flow of irrigant solution throughout the canal.
  Finally, the canal was rinsed with sterile water using a syringe with a side-vented 30 G needle 1 mm shorter than the working length. A second sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect the presence of blood and the millimeters of blood inside the root canal was measured again according the previous criteria.
  Arms: Control

SUMMARY:
The persistence of blood may significantly affect final sealing with the persistence of microleakage (Zmener et al. 2008, Roggendorf et al. 2007).

In cases of copious bleeding from root canals, calcium hydroxide, anesthetic solution with 1:50,000 epinephrine or ferric sulfate placed on a sterile paper cone, are recognized as effective hemostatic agents (Magnusson 1971, Kouri et al. 1969, Dannenberg 1974).

The purpose of this study was to test the reduction of root canal bleeding in terms of significant percentage change for millimeters of blood in the canal at 2 different time points (baseline and after treatment with HybenX )

DETAILED DESCRIPTION:
A new device (HYBENX®, EPIEN Medical, Saint Paul, MN, USA) has been developed with the purpose of destroying dental biofilm. The material is a mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%).

This device has been successfully used in periodontology. Recent studies (Pini-Prato et al. 2016a, Isola et al. 2017) have demonstrated the effectiveness of the oral tissue decontaminant material in the treatment of clinical cases showing acute periodontal abscess without the use of systemic or local antibiotics. Similar favorable effects were obtained in the treatment of peri-implant mucositis and peri-implantitis (Pini-Prato et al. 2016b, Lopez et al. 2016). In addition, a randomized controlled trial (RCT) also demonstrated beneficial effects of the material in the treatment of oral aphthae (Porter et al. 2009).

Based on this scientific information, a clinical and microbiological study has been planned using the decontaminant device in cases of teeth with necrotic pulp with the aim to destroy the dental biofilm of root canals. The ability of the decontaminant device to immediately stop bleeding during canal instrumentation was found out accidentally during the procedures of this still unpublished trial.

Due to this fact, the authors were interested in evaluating the coagulation property of the material. The purpose of this study was to test the reduction of root canal bleeding in terms of significant percentage change for millimeters of blood in the canal at 2 different time points (before and after treatment with HybenX ) A single center, participants and data analyst blind, two-arm, randomized, placebo controlled clinical trial study was performed following the CONSORT statement in the Endodontics Department, University Hospital Florence Careggi, Florence, Italy.

The study population consisted of patients that were treated by Endodontics Department of the University Hospital of Florence Careggi, Italy. Subject inclusion criteria were: patients aged between 20 and 60 years, able and willing to sign a consent form, single-rooted teeth with necrotic pulp confirmed by electric vitality test, associated with healthy periodontium, physiologic sulcus depth (<3 mm), and absence of bleeding on probing of the involved teeth.

Exclusion criteria were: patients with systemic diseases using anticoagulants, antibiotics, or anti-inflammatory therapies in the last 30 days, patients with allergy to sulfur in any form, and pregnancy. All subjects were informed of the nature and potential risks and benefits of their participation in the study. They also received information on the duration of the procedure, and the possible intraoperative and postoperative complications.

Treatment The root canal therapy procedure was standardized and limited to one experienced endodontist (R.P.). Treatments were performed at the Endodontics Departments of the University Hospital of Florence Careggi, Italy, under local anesthesia using 1.8 mL mepivacaine hydrochloride (Optocaine; Molteni Dental SRL, Scandicci, Italy), and the teeth were isolated with rubber dams. After preparing the access cavity, the working length was determined with an electronic apex locator (Propex II Dentsply Maillefer Instruments, Ballaigues, Switzerland) with a size 10 k-file. Root canals were shaped using ProTaper Universal NiTi files (Dentsply Maillefer Instruments, Ballaigues, Switzerland) in the following sequence: S1, S2, F1, F2, F3 until each instrument reached the working length. After each instrument, the root canals were rinsed with NaClO (Niclor 5, Ogna, Italy) using a syringe with a side-vented 30 G needle. ProTaper NiTi instruments were driven with an endodontic motor (XSmart Endo Motor, Dentsply Maillefer Instruments, Ballaigues, Switzerland) with a 16:1 contrangle set up as suggested by the manufacturer.

After the root canal, shaping was performed, and a first sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect blood presence.

With a caliber, on the sterile paper cone, the millimeters of blood present within the root canal were measured.

Only the teeth that at this point showed 1 or more millimeters of blood within the root canal were included in the present study and randomized to the two experimental groups.

Before further treatment, the teeth were allocated to an experimental (HybenX) or a control group (sterile saline solution) according to an uneven block randomization designed by the statistician (A.N.). For each tooth, a closed envelope was opened in a consecutive order, assigning the tooth to either the experimental or the control group HybenX was approved as a Class I CE medical device by the Italian Ministry of Health (no. 483768) on February 7, 2012.

HybenX Group The material was introduced inside the root canal using the pre-dosed syringe for 20 seconds with a sterile paper point with and up and down movement up to the working length.

Finally, the canal was rinsed with sterile water using a syringe with a side-vented 30 G needle 1 mm shorter than the working length.

A second sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect the presence of blood and the millimeters of blood inside the root canal was measured again according the previous criteria.

Statistical Analysis Data were analyzed using SAS Version 9.3 software (SAS Institute, Inc., Cary, NC). A preliminary Levene's test was performed to verify the homogeneity of variance for the percentage change in the two groups.

Since the two groups showed homogeneity of the variance a t-test was performed to verify the null hypothesis by using a type I error equal to 0.05.

In order to confirm the firmness of the results a Wilcoxon non-parametric test was also carried out.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20 and 60 years
* patients able and willing to sign a consent form,
* single-rooted teeth with necrotic pulp confirmed by electric vitality test
* healthy periodontium
* physiologic sulcus depth (<3 mm)
* absence of bleeding on probing of the involved teeth.

Exclusion Criteria:

* patients with systemic diseases
* patients using anticoagulants in the last 30 days
* patients using antibiotics in the last 30 days
* patients using anti-inflammatory therapies in the last 30 days
* patients with allergy to sulfur in any form
* pregnancy.

All subjects were informed of the nature and potential risks and benefits of their participation in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AOUCareggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pini-Prato G, Magnani C, Rotundo R. Nonsurgical Treatment of Peri-implantitis Using the Biofilm Decontamination Approach: A Case Report Study. Int J Periodontics Restorative Dent. 2016 May-Jun;36(3):383-91. doi: 10.11607/prd.2653. PMID 27100808
- [Background] Lopez MA, Andreasi Bassi M, Confalone L, Silvestre F, Arcuri C. The treatment of peri-implant diseases: a new approach using hybenx(R) as a decontaminant for implant surface and oral tissues. Oral Implantol (Rome). 2016 Nov 13;9(3):106-114. doi: 10.11138/orl/2016.9.3.106. eCollection 2016 Jul-Sep. PMID 28042438
- [Background] Porter SR, Al-Johani K, Fedele S, Moles DR. Randomised controlled trial of the efficacy of HybenX in the symptomatic treatment of recurrent aphthous stomatitis. Oral Dis. 2009 Mar;15(2):155-61. doi: 10.1111/j.1601-0825.2008.01503.x. PMID 19207485
- [Background] Zmener O, Pameijer CH, Serrano SA, Vidueira M, Macchi RL. Significance of moist root canal dentin with the use of methacrylate-based endodontic sealers: an in vitro coronal dye leakage study. J Endod. 2008 Jan;34(1):76-9. doi: 10.1016/j.joen.2007.10.012. PMID 18155498
- [Background] Roggendorf MJ, Ebert J, Petschelt A, Frankenberger R. Influence of moisture on the apical seal of root canal fillings with five different types of sealer. J Endod. 2007 Jan;33(1):31-3. doi: 10.1016/j.joen.2006.07.006. Epub 2006 Oct 13. PMID 17185125
- [Background] Magnusson B. Therapeutic pulpotomy in primary molars--clinical and histological follow-up. II. Zinc oxide-eugenol as wound dressing. Odontol Revy. 1971;22(1):45-54. No abstract available. PMID 5280515
- [Background] Kouri EM, Matthews JL, Taylor PP. Epinephrine in pulpotomy. ASDC J Dent Child. 1969 Mar-Apr;36(2):123-8. No abstract available. PMID 4888301
- [Background] Dannenberg JL. Pedodontic endodontics. Dent Clin North Am. 1974 Apr;18(2):367-77. No abstract available. PMID 4274315
- [Background] Isola G, Matarese G, Williams RC, Siciliano VI, Alibrandi A, Cordasco G, Ramaglia L. The effects of a desiccant agent in the treatment of chronic periodontitis: a randomized, controlled clinical trial. Clin Oral Investig. 2018 Mar;22(2):791-800. doi: 10.1007/s00784-017-2154-7. Epub 2017 Jun 17. PMID 28624914
- [Background] Pini-Prato G, Magnani C, Rotundo R. Treatment of Acute Periodontal Abscesses Using the Biofilm Decontamination Approach: A Case Report Study. Int J Periodontics Restorative Dent. 2016 Jan-Feb;36(1):55-63. doi: 10.11607/prd.2557. PMID 26697553

RESULTS

PARTICIPANT FLOW:
Groups:
- HybenX ®: 1 cc of mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%) for 20 sec
  HybenX: The material was introduced inside the root canal using the pre-dosed syringe for 20 seconds with a sterile paper point with and up and down movement up to the working length.
  Finally, the canal was rinsed with sterile water using a syringe with a side-vented 30 G needle 1 mm shorter than the working length.
  A second sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect the presence of blood and the millimeters of blood inside the root canal was measured again according the previous criteria.
- Control: 5 cc of sterile saline water for 20 sec
  Placebo control: The root canal was irrigated with sterile saline water with a syringe and a side-vented 30G needle activated for 20 seconds with a sterile paper point with and up and down movement up to the working length to ensure a flow of irrigant solution throughout the canal.
  Finally, the canal was rinsed with sterile water using a syringe with a side-vented 30 G needle 1 mm shorter than the working length. A second sterile paper point was introduced in the root canal, up to the working length, for 10 seconds to detect the presence of blood and the millimeters of blood inside the root canal was measured again according the previous criteria.
Period: Overall Study
Arm/Group | HybenX ® | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HybenX ® | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (9.9) | 35.2 (10.2) | 37.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Root Canal Bleeding
Description: After the root canal, shaping was performed a first sterile paper point was introduced in the root canal, up to the working length, to detect blood presence.
  The millimeters of blood on the paper point were measured with a caliber. After the intervention (HybenX or placebo) a second sterile paper point was introduced in the root canal, up to the working length, to detect the presence of blood according the previous criteria
Time Frame: Baseline and After Treatment (20 seconds)
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: teeth
Arm/Group | HybenX ® | Control
Number analyzed (Participants) | 30 | 30
Number analyzed (teeth) | 30 | 30
millimeters
  Baseline | 3.40 (1.54) | 3.73 (1.14)
  After treatment | 0.26 (0.69) | 3.03 (1.30)
Statistical Analysis 1: Comparison: HybenX ® vs Control; Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [0.66 to 0.82]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | HybenX ® | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03336853/Prot_SAP_001.pdf